CLINICAL TRIAL: NCT06352944
Title: Bronchoscopic Derived Bronchoalveolar Lavage Procalcitonin as a Marker of Severity of Non-cystic Fibrosis Bronchiectasis in Children
Brief Title: Procalcitonin as a Marker of Severity of Non-cystic Fibrosis Bronchiectasis in Children
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Maram Mohamed Amir Fathy, assistant lecturer, Assiut University
Other Study IDs: AssiutMD
Record Dates: First submitted 2024-04-03; First posted 2024-04-08 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Non-cystic Fibrosis Bronchiectasis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Diagnostic Test: procalcitonin — level of procalcitonin in bronchoalveolar lavage

SUMMARY:
The aim of this study is to evaluate the role of procalcitonin in bronchoalveolar lavage as a biomarker for assessment of severity of non-CF bronchiectasis in children in correlation with other markers (functional and radiological severity )

DETAILED DESCRIPTION:
• The severity of bronchiectasis will be assessed using forced expiratory volume in 1s (FEV1), and bronchiectasis severity scores which included bronchiectasis severity index (BSI) , FEV1, chronic colonization, extension of lobes and dyspnea which were performed to assess non-CF bronchiectasis patients.

BSI score

* This score incorporates 9 variables. The total score is calculated by summing the scores for each variable and can range from 0 to 26 points. According to the overall score, patients are classified into three classes: patients with low BSI score (0---4 points), intermediate BSI score (5---8 points), high BSI score (≥9 points)
* chest X ray and HRCT of the chest: to assess the radiological severity of bronchiectasis using the radiological findings will be measured by assessing the most recent chest X ray and HRCT of the chest performed in the last six months using Bhalla score(10)
* Culture and sensitivity from bronchoalveolar lavage for isolation of pseudomonas aeruginosa and any other organism.
* Sputum procalcitonin level was measured in BAL samples using bronchoscopy.
* Bronchoscopy: would be undertaken when the children were in a stable clinical condition as part of their annual review

ELIGIBILITY:
Inclusion Criteria:

1. Children of both sex
2. Children aged from 6-17 years old.
3. Documented diagnosis of non-CF bronchiectasis by confirmed bronchiectasis findings using high-resolution computed tomographic (HRCT) lung scanning, and clinical symptoms consistent with bronchiectasis with a negative sweat test

Exclusion Criteria:

1. Age less than 6 years or more than 17 years.
2. Children Diagnosed with cystic fibrosis bronchiectasis with confirmed positive sweat chloride test(6).
3. If there was a history of a recent exacerbation during the previous month preceding the study.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children aged from 6 to 18 years diagnosed with Non-cystic fibrosis bronchiectasis
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
procalcitonin level in bronchoalveolar lavage as a biomarker for assessment of severity of non-CF bronchiectasis in children | 2 years
  comparison between procalcitonin level in Bronchoalveolar lavage and other markers of severity of bronchiectasis

CONTACTS AND LOCATIONS:
Overall Officials: Yasser F abdelrahem, professor, Study Director — Assiut University

IPD SHARING:
Plan to Share IPD: No